CLINICAL TRIAL: NCT04416074
Title: An Online 5-week Professional Identity Group Psychotherapy for Nursing Student During Clinical Rotation Practice
Brief Title: An Online 5-week Professional Identity Group Psychotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central South University (Other)
Collaborators: Fudan University (Other)
Responsible Party: Principal Investigator, Anni Wang, Principal Investigator, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5-week Identity intervention
Record Dates: First submitted 2020-05-30; First posted 2020-06-04 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-05

CONDITIONS: Identification (Psychology)
Keywords: Professional identity; Career self-efficacy; Resilience

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group psychotherapy group (Experimental): Students will be intervened by an online 5-week professional identity group psychotherapy.
  Interventions: Behavioral: An online 5-week professional identity group psychotherapy
- Controlled message push group (Other): Students will receive online messages of self-care knowledge forward by researchers.
  Interventions: Other: Message push

INTERVENTIONS:
Behavioral: An online 5-week professional identity group psychotherapy — This is an online 5-week group psychological intervention for the nursing students during clinical rotation practice. It aims at promoting the professional identity and career sefl-efficacy for them. There are five sessions in the intervention, and each session lasts from 60min to 90min at each week. The intervention will be delivered via an online meeting software, like Zoom. There will be 15-20 students in one meeting group.
  Arms: Group psychotherapy group
Other: Message push — Controlled group will receive online messages of self-care knowledge forward by researchers once per week. The knowledge contain stress regulation, strategies for relaxation, self-protection during clinical practice.
  Arms: Controlled message push group

SUMMARY:
This is an online 5-week group psychological intervention for the nursing students during clinical rotation practice. It aims at promoting the professional identity and career sefl-efficacy for them.

DETAILED DESCRIPTION:
Those 110 participants come from two classes in the same grade. One will be randomly allocated as the intervention group, the other will be control group. The intervention will be delivered via an online meeting software, like Zoom. The control group will received five messages fo self care messages forward by the researcher.

ELIGIBILITY:
Inclusion Criteria:

* Full time nursing student
* During clinical rotation practice
* Able to comprehend the intervention

Exclusion Criteria:

* Visual impairment
* Absent more than twice of the intervention

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 110 (Actual)
Dates: Start 2020-05-10 (Actual); Primary Completion 2020-06-13 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
Professional identity | We will measure the score of professional identity before intervention and immediately after intervention.
  Professional identity in recent one week measured by Chinese Profession identity scale for nursing student, ranging from 17 to 85, with higher score reflects higher level of idnetity.
Career self-efficacy | We will measure the score of career self-efficacy before intervention and immediately after intervention.
  Career self-efficacy in recent one week measured by the Chinese career self-efficacy scale for nursing student, ranging from 27-135, with higher score reflects higher level of career self-efficacy.

SECONDARY OUTCOMES:
Stress | We will measure the score of stress before intervention and immediately after intervention.
  A reflection of one's perceived stress in recent month measured by the subscale from the Depression, Anxiety, and Stress Scale (DASS-21). The score rangs from 0-21, with higher score reflects higher level of stress.
Resilience | We will measure the score of resilience before intervention and immediately after intervention.
  Resilience in recent one week measured by the Chinese version of Connor-Davidson Resilience Scale-10. The score ranges from 0-40, with higher score reflects higher level of resilience.

OTHER OUTCOMES:
General rating | We will measure this immediately after intervention.
  Several descriptive question to gather the feedback of the intervention. Each question will be rated from 0 to 5, with higher score reflects higher level of satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Anni Wang, Dr., Principal Investigator — School of Nursing, Fudan University
Locations (1):
- School of Nursing, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
The participants are not willing to share the data.

REFERENCES:
- [Background] Ohlen J, Segesten K. The professional identity of the nurse: concept analysis and development. J Adv Nurs. 1998 Oct;28(4):720-7. doi: 10.1046/j.1365-2648.1998.00704.x. PMID 9829659
- [Background] Kirpal, S.J.C.D.I., Work identities of nurses: Between caring and efficiency demands. 2004.
- [Background] Roberts SJ. Development of a positive professional identity: liberating oneself from the oppressor within. ANS Adv Nurs Sci. 2000 Jun;22(4):71-82. doi: 10.1097/00012272-200006000-00007. PMID 10852670
- [Background] Megginson LA. RN-BSN education: 21st century barriers and incentives. J Nurs Manag. 2008 Jan;16(1):47-55. doi: 10.1111/j.1365-2934.2007.00784.x. PMID 18211335
- [Background] Cook TH, Gilmer MJ, Bess CJ. Beginning students' definitions of nursing: an inductive framework of professional identity. J Nurs Educ. 2003 Jul;42(7):311-7. doi: 10.3928/0148-4834-20030701-08. PMID 12873061
- [Background] Hunter B, Segrott J. Re-mapping client journeys and professional identities: a review of the literature on clinical pathways. Int J Nurs Stud. 2008 Apr;45(4):608-25. doi: 10.1016/j.ijnurstu.2007.04.001. Epub 2007 May 23. PMID 17524406
- [Background] Yamagishi M, Kobayashi T, Nakamura Y. Effects of web-based career identity training for stress management among Japanese nurses: a randomized control trial. J Occup Health. 2008;50(2):191-3. doi: 10.1539/joh.l7086. No abstract available. PMID 18403870
- [Derived] Kunzler AM, Helmreich I, Konig J, Chmitorz A, Wessa M, Binder H, Lieb K. Psychological interventions to foster resilience in healthcare students. Cochrane Database Syst Rev. 2020 Jul 20;7(7):CD013684. doi: 10.1002/14651858.CD013684. PMID 32691879

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-03): https://cdn.clinicaltrials.gov/large-docs/74/NCT04416074/Prot_SAP_000.pdf